CLINICAL TRIAL: NCT03816735
Title: Erbium:Yag Laser vs Hyaluronic Acid Suppository for GSM in Breast Cancer (BC)
Brief Title: Laser vs Hyaluronic Acid for GSM in Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30-225 ex 17/18
Record Dates: First submitted 2019-01-23; First posted 2019-01-25 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Urogenital Disease
MeSH Terms: conditions — Urogenital Diseases

STUDY DESIGN:
Intervention Model Description: Randomized open study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- hyaluronic acid suppository therapy (Active Comparator): Women receive a vaginal suppository called "Cikatridina" manufactured by the company Angelini to treat women with GSM. Angelini Pharma Österreich GmbH's headquarters are located in Brigittenauer Lände 50-54, 1200 Wien, Austria. The suppositories contain ontain hyaluronic acid, tea tree oil, tigergras extract, and aloe vera.
  Interventions: Device: Cikatridina
- Juliet feminine laser (Active Comparator): The fractional microablative laser with 2940 nm wavelength has a high degree of absorption in water and selectively stimulates the synthesis of sub-mucosal collagen. The erbium-doped yttrium-aluminum-garnet (Er:YAG) laser has been successfully used in the field of plastic skin rejuvenation and reconstruction. The procedure is based on photothermic treatment of connective tissue: It has been established in animal and human studies that it affects collagen remodeling resulting in tightening of the supportive tissue.
  Interventions: Device: Juliet Feminine Laser

INTERVENTIONS:
Device: Cikatridina — Women are asked to insert the suppositories according to the manufacturer's protocol.
  Arms: hyaluronic acid suppository therapy
Device: Juliet Feminine Laser — Women will receive the laser treatment twice during the study period.
  Arms: Juliet feminine laser

SUMMARY:
All women from the outpatient department with a history of BC and GSM (genitourinary symptoms of menopause) symptoms will be invited to participate.

After informed consent patients are either randomized to intravaginal laser or hyaluronic acid suppository treatment intravaginally, respectively. Laser treatment will be performed twice, at baseline and after 1 month. The intravaginal hyaluronic acid suppository therapy will be applied daily during the first 10 days and then every third day until the three months follow-up.

At baseline and three months follow-up the following questionnaires will be filled out (VAS, (PGI-I, PGI-S, Female Sexual health questionnaire (EORTC), Baessler questionnaire, EORTC quality of life questionnaire, ZUF-8).

DETAILED DESCRIPTION:
Device I- Laser The laser device is the Juliet feminine laser to treat women with SUI (Stress Urinary Incontinence), GSM and vaginal laxity. Asclepion' s headquarters are located in "Asclepion Laser Technologies GmbH - Brüsseler Str. 10 - 07747 Jena - Germany".

Device II- Suppository The second device is a vaginal suppository called "Cikatridina" manufactured by the company Angelini to treat women with GSM. Angelini Pharma Österreich GmbH's headquarters are located in Brigittenauer Lände 50-54, 1200 Wien, Austria.

ELIGIBILITY:
Inclusion criteria

* genital symptoms of dryness/ burning/ irritation

  * and/ or lack of lubrication during sexual intercourse/ sexual discomfort or pain
  * and/or symptoms of urgency and dysuria or recurrent urinary tract infection
* Age 18-80
* History of BC and/ or DCIS
* Completed locoregional therapy
* Current antihormonal therapy for BC possible
* Intravaginal treatment with creams/ suppositories other than study medicationshould be ceased during the trial

Exclusion criteria:

* Current or past genitourinary malignancy
* Abnormal PAP smear
* Current genitourinary tract infection
* Abnormal uterine bleeding
* photosensitive medication

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2019-01-24 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
genitorurinary symptoms of menopause (GSM) determined by vaginal health index score | 3 months
  Vaginal Health Score Index (VHIS) evaluates the appearance of the vaginal mucosa (elasticity, pH, vaginal discharge, mucosal integrity and moisture) on a scale from 1 to 5 each. The lower the score the worse the symptom.

SECONDARY OUTCOMES:
Symptoms severity- visual analogue scale | 3 months
  A visual analogue scale (VAS) is used for assessment for the subjective bother of GSM. The lower the score the less bothering are the symptoms.
Treatment discomfort / pain; assessed by visual analogue scale | 3 months
  At the end of each laser treatment session or at 3 months for the vaginal suppository group patients are asked to indicate the degree of discomfort or pain during laser therapy/vaginal insertion of the suppositories on a scale ranging from 0 (no discomfort/pain) to 10 (worst possible discomfort/pain)
Patient Global Impression of Improvement | 3 months
  The Patient Global Impression of Improvement (PGI-I) are robust and valid instruments to assess disease severity, bother and improvement after treatment in women. It ranges from very much improved to a lot worse on 7 likert scale.
Patient Global Impression of Severity | 3 months
  The Patient Global Impression of Severity (PGI-S) is a global index that may be used to rate the severity of a specific condition (a single-state scale). The PGI scales are robust and valid instruments to assess disease severity, bother and improvement after treatment. The patient can choose from 4 answers including none, mild, moderate and severe.
Female Sexual health | 3 months
  The Female Sexual health is assessed with the European Organisation for Research and Treatment of Cancer (EORTC) sexual health questionnaire and is a validated questionnaire which assesses physical, psychological, and social aspects of sexuality of cancer survivors. It is a 22 item questionnaire.The higher the score the better is the sexual function.
pelvic floor symptoms | 3 months
  A validated self-administered pelvic floor questionnaire (Baessler) will be used to assess urogentinal symptoms. Questions regarding bladder (15), bowel (12), and sexual function (10), and pelvic organ prolapse symptoms (five) are grouped according to the physiological functions of the pelvic floor: bladder function, bowel function, prolapse symptoms, and sexual function domains. Quality of life measures and bothersomeness ratings were integrated into the four domains. Frequency, severity, and bothersomeness of pelvic floor symptoms are assessed using a four-point scoring system for most items in the questionnaire, apart from defecation frequency, bowel consistency, sufficient lubrication, and the reason for sexual abstinence. The lower the score the less pelvic floor symptoms the patients have.
Patient satisfaction with treatment/ inpatient management | 3 months
  "Fragebogen zur Patientenzufriedenheit - ZUF8". The questionnaire, the German version of the original "Client Satisfaction Questionnaire-CSQ8", is a validated tool for measuring global patient satisfaction at the end of inpatient treatment. The Zuf-8 is an 8-items questionnaire to assess satisfaction in patients undergoing inpatient treatment. At 3 months treatment satisfaction will be assessed using an adopted version of the questionnaire. The lower the score the higher is the patient satiscation.
Discontinuation rate | 3 months
  Number of patients who discontinue treatment
Dyspareunia rate | 3 months
  evaluated by a single item of the Baessler questionnaire. The rate will be given in number and percent.
Quality of life: EORTC quality of life questionnaire | 3 months
  Determined by the European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire. The questionnaire is a 47 item questionnaire and assess quality of life. The lower the score the better the quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics, Medical University Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gold D, Nicolay L, Avian A, Greimel E, Balic M, Pristauz-Telsnigg G, Tamussino K, Trutnovsky G. Vaginal laser therapy versus hyaluronic acid suppositories for women with symptoms of urogenital atrophy after treatment for breast cancer: A randomized controlled trial. Maturitas. 2023 Jan;167:1-7. doi: 10.1016/j.maturitas.2022.08.013. Epub 2022 Sep 9. PMID 36279690
- [Derived] European Urogynaecological Association 2021 Annual Meeting | Hybrid Edition. Female Pelvic Med Reconstr Surg. 2022 Apr 1;28(4):244-271. doi: 10.1097/SPV.0000000000001172. No abstract available. PMID 35443258